CLINICAL TRIAL: NCT00002305
Title: Multicenter Comparison of Fluconazole (UK-49,858) and Amphotericin B as Treatment for Acute Cryptococcal Meningitis
Brief Title: A Comparison of Fluconazole and Amphotericin B in the Treatment of Cryptococcal Meningitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 012F; 056-159
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-12

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Drug Therapy, Combination; Fluconazole; Flucytosine; Acquired Immunodeficiency Syndrome; Amphotericin B
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Acquired Immunodeficiency Syndrome | interventions — Flucytosine; Fluconazole; Amphotericin B

INTERVENTIONS:
Drug: Flucytosine
Drug: Fluconazole
Drug: Amphotericin B

SUMMARY:
To compare the safety and effectiveness of fluconazole and amphotericin B, alone or in combination with flucytosine, as treatment for acute cryptococcal meningitis.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Immunosuppressant therapy.
* Antiviral therapy such as zidovudine.
* Prophylaxis for Pneumocystis carinii pneumonia.

Concurrent Treatment:

Allowed:

* Radiation therapy for mucocutaneous Kaposi's sarcoma.

Written informed consent must be obtained for each patient, either from the patient himself or from the patient's legal guardian.

* No prior systemic antifungal therapy for cryptococcosis.
* Relapse after prior therapy.
* Success of prior therapy must have been documented by negative cerebrospinal fluid (CSF) culture at the end of therapy. Following prior therapy, such patients may not have received more than 1 mg/kg/wk amphotericin B in the 4 weeks before entry into study.

Prior Medication:

Allowed:

* Immunosuppressant therapy.
* Antiviral therapy (such as zidovudine).
* Prophylaxis for Pneumocystis carinii pneumonia.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Evidence of acute or chronic meningitis based upon any etiology other than cryptococcosis.
* History of allergy to or intolerance of imidazoles, azoles, or amphotericin B.
* Moderate or severe liver disease.
* Comatose.
* Unlikely to survive more than 2 weeks.
* Any exceptions to these prohibitions of concomitant medications must be approved by Pfizer Central Research.

Concurrent Medication:

Excluded:

* Coumadin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Phenytoin.
* Immunostimulants.
* Investigational drugs or approved (licensed) drugs for investigational indications.
* Any exceptions to these prohibitions of concomitant medications must be approved by Pfizer Central Research.
* Excluded within 4 weeks of study entry:
* Greater than 1 mg/kg/wk amphotericin B.

Concurrent Treatment:

Excluded:

* Lymphocyte replacement.

Patients with the following are excluded:

* Evidence of acute or chronic meningitis based upon any etiology other than cryptococcosis.
* History of allergy to or intolerance of imidazoles, azoles, or amphotericin B.
* Moderate or severe liver disease.
* Comatose.
* Unlikely to survive more than 2 weeks.

Prior Medication:

Excluded:

* Coumadin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Phenytoin.
* Immunostimulants.
* Investigational drugs or approved (licensed) drugs for investigational indications.
* Excluded within 4 weeks of study entry:
* Greater than 1 mg/kg/wk amphotericin B.

Prior Treatment:

Excluded:

* Lymphocyte replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (45):
- United States (44):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Tucson Veterans Administration Med Ctr, Tucson, Arizona
  - UCLA CARE Ctr, Los Angeles, California
  - Dr Shelly Gordon, San Francisco, California
  - Dr Martin Mass, San Francisco, California
  - Dr Paul Rothman, Sherman Oaks, California
  - Christiana Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Univ of South Florida, Tampa, Florida
  - Emory Univ School of Medicine, Atlanta, Georgia
  - Med College of Georgia, Augusta, Georgia
  - DeKalb Gen Hosp, Decatur, Georgia
  - Northwestern Univ Med School, Chicago, Illinois
  - Louisiana State Univ School of Medicine, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Dr Michael Bach, Portland, Maine
  - Univ of Maryland / Inst of Human Virology, Baltimore, Maryland
  - Loch Raven Veterans Hosp, Baltimore, Maryland
  - New England Med Ctr, Boston, Massachusetts
  - Univ Hosp, Boston, Massachusetts
  - Ann Arbor Veterans Administration Med Ctr, Ann Arbor, Michigan
  - Harper Hosp, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Washington Univ School of Medicine, St Louis, Missouri
  - Albany Med College / AIDS Treatment Ctr, Albany, New York
  - Jewish Hosp Ctr Affiliation, Jamaica, New York
  - Chelsea Village Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Columbia Univ, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Univ of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Cincinnati Veterans Adm Med Ctr / Univ Hosp, Cincinnati, Ohio
  - Ohio State Univ Hosp, Columbus, Ohio
  - Univ of Tennessee, Memphis, Tennessee
  - Dr Daniel Barbaro, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - United States Air Force Med Ctr, Lackland Air Force Base, Texas
  - Univ TX San Antonio Health Science Ctr, San Antonio, Texas
  - Richmond AIDS Consortium, Richmond, Virginia
  - CHG-118 Group Health / Cooperative of Puget Sound, Seattle, Washington
- Saint Michael's Hosp, Toronto, Ontario, Canada